CLINICAL TRIAL: NCT02949609
Title: Mirror Therapy: Effects on Functional Recuperation of Severe Upper Limb Paresis After Stroke
Acronym: MT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: investigator
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Leemann Beatrice, Medical Doctor (MD), University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-00091
Record Dates: First submitted 2016-10-25; First posted 2016-10-31 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Stroke
Keywords: stroke; mirror therapy; neurorehabilitation
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mirror Therapy (MT) (Experimental): Standard therapy + 30 min/day of mirror therapy, 5 days/week, for 4 weeks, administered by experienced physical and occupational therapists.
  Interventions: Other: Mirror Therapy
- Control Therapy (CT) (Active Comparator): Standard therapy + 30 min/day of CT.
  Interventions: Other: Control Therapy

INTERVENTIONS:
Other: Mirror Therapy — Mirror therapy will consist in placing a large mirror in the sagittal plane of the subject so as to reflect his healthy arm while hiding the paretic one, and then asking him to perform movements of his healthy arm while looking at its reflection in the mirror.
  Arms: Mirror Therapy (MT)
Other: Control Therapy — Performance of the same movements as the experimental group without the mirror or instructions as to where to look, 5 days/week, for 4 weeks.
  Arms: Control Therapy (CT)

SUMMARY:
After stroke, patients frequently suffer from arm or hand weakness. There are numerous rehabilitation methods to stimulate recovery, amongst which mirror therapy (MT). It is particularly interesting in cases for which impairment is severe, as many other forms of therapy are often impossible.

During MT, a mirror is placed in the midsagittal plane, so as to hide the impaired limb. Thereafter, the subject is asked to move his unimpaired limb while looking at its reflection in the mirror, thereby creating the illusion that the contralateral, impaired limb is moving.

The objective of this study is to better determine the efficacy of MT. The investigators will therefore compare recovery of arm function in two groups of patient, that perform a regimen of 30 minutes of therapy, 5 times a week, for 4 weeks on top of conventional therapy. One group performs MT and the other one performs a therapy in which the same movements are performed, but without the use of a mirror, with unrestricted view of both limbs. Allocation to each group will be randomized. Arm function will be evaluated by use of a scale before, during and after the 4 week period. The assessor for the primary outcome measure will not know in which group the patient is. There will be a total of 30 patients included over a one year study period.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke, diagnosed clinically and by imagery, more than one month after onset;
* Severe upper limb paresis with Upper-Extremity Fugl-Meyer Score < 19/60 .

Exclusion Criteria:

* Significant limitation in upper limb function predating the recent stroke, caused by former symptomatic stroke and/or an orthopedic/rheumatologic disease;
* Neuropsychologic or psychiatric impairment with significant interference with participation in therapy;
* Severe visual impairment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-06-17; Primary Completion 2017-11-17 (Actual); Study Completion 2017-11-17 (Actual)

PRIMARY OUTCOMES:
Change in Fugl Meyer Assessment - Upper Limb (FMA-UE) | Baseline, 2 weeks and 4 weeks after start of therapy. Additional follow-up visit min. 6 weeks after discharge from rehabilitation.
  Change in Fugl Meyer Assessment - Upper Limb (FMA-UE) at different time points: before, during, after intervention and after a 6 week follow-up.

SECONDARY OUTCOMES:
Change in Functional Independence Measure (FIM) | Baseline, 2 weeks and 4 weeks after start of therapy. Additional follow-up visit min. 6 weeks after discharge from rehabilitation.
  Change in Functional Independence Measure (FIM) at different time points: before, during, after intervention and after a 6 week follow-up.
Change in Bell cancellation task | Baseline, 2 weeks and 4 weeks after start of therapy. Additional follow-up visit min. 6 weeks after discharge from rehabilitation.
  Change in Bell cancellation task at different time points: before, during, after intervention and after a 6 week follow-up.
Change in Line bisection task | Baseline, 2 weeks and 4 weeks after start of therapy. Additional follow-up visit min. 6 weeks after discharge from rehabilitation.
  Change in Line bisection task at different time points: before, during, after intervention and after a 6 week follow-up.
Change in Numeric pain scale | Baseline, 2 weeks and 4 weeks after start of therapy. Additional follow-up visit min. 6 weeks after discharge from rehabilitation.
  Change in Numeric pain scale at different time points: before, during, after intervention and after a 6 week follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice Leemann, Doctor, Principal Investigator — University Hospital, Geneva
Locations (1):
- Service de Neurorééducation - Hôpitaux Universitaires de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No